CLINICAL TRIAL: NCT05010044
Title: Mindfulness-based Cognitive Therapy for Psoriasis Patients With Anxiety and Depression
Brief Title: MBCT for Psoriasis Patients With Anxiety and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2019-027
Record Dates: First submitted 2021-07-14; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants received MBCT once a week for 8 weeks (Experimental): Participants received MBCT once a week for 8 weeks. At the same time, the drug therapy for psoriasis was used .
  Interventions: Behavioral: mindfulness-based cognitive therapy (MBCT); Other: Antipsoriatic treatment
- Active comparator (Active Comparator): Only the drug therapy for psoriasis was used .
  Interventions: Other: Antipsoriatic treatment

INTERVENTIONS:
Behavioral: mindfulness-based cognitive therapy (MBCT) — Mindfulness- Based Cognitive Therapy (MBCT) It involves practicing to be present 'in the moment' and an attitude of non- judgmental acceptance with the aim to maintain awareness, disengaging oneself from strong attachment and thereby developing a greater sense of emotional balance and well-being.
  Arms: Participants received MBCT once a week for 8 weeks
Other: Antipsoriatic treatment — The routine drug therapy for psoriasis.

SUMMARY:
This study investigates the effectiveness of a 24-week mindfulness intervention in reducing symptoms in psoriasis patients with anxiety and depression.

DETAILED DESCRIPTION:
An adapted MBCT intervention will be offered to people with psoriasis with depression and/or anxiety. 8-week long MBCT therapy will be held between August 2021 and Jan 2022, based on the adapted protocol. The MBCT intervention will consist of 30-minute weekly groups focused on teaching mindfulness techniques and ways to recognize cognitive patterns that can increase anxiety and/or depression. Participants will be recruited from the community, according to the eligibility criteria detailed below. For all participants, anxiety and/or depressive symptom severity(SAS/SDS), PASI,DLQI,(as measured with standardized, validated scales) will be compared baseline and weeks 2;4;8;12;16;20;24. Itch intensity ,itch perception ,quality of sleep, hours missing at work ,helpfulness of common itch therapies serve as the secondary outcome, using a paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* the age ranged from 18 to 70 years old
* fulfilled the Classification Criteria for Psoriasis
* the score of the SDS > 50 and / or SAS >50
* Participant has normal or corrected to normal vision and hearing
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Participant has insufficient manual dexterity for the computerized tasks
* severe systemic diseases
* patients with severe mental illness or taking psychotic drugs
* Pregnancy
* No access to the internet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on the Psoriasis Area and Severity Index (PASI) | Baseline and Week 2;4;8;12;16;20;24
  PASI a measurement that combines severity of lesions and the area affected in one score that ranges from 0 to 72 .
Change from Baseline on the Dermatology Life Quality Index (DLQI) | Baseline and Week 2;4;8;12;16;20;24
  The DLQI is a 10-item questionnaire measuring the effect of dermatological diseases on patients over the last week. The DLQI total score is the sum of each individual item score and ranges from 0 or 1 to 30 .
Change from Baseline on the Self-rating Depression Scale (SDS) | Baseline and Week 2;4;8;12;16;20;24
  In the main component of the SDS , patients are asked 20 questions about Mental and physical feelings of emotional experience, and the patients determine the quality of emotion by selecting one of the options: Occasionally=1, sometimes=2, often=3, and continuously=4.
Change from Baseline on the Self-rating Anxiety Scale (SAS). | Baseline and Week 2;4;8;12;16;20;24
  In the main component of the SAS , patients are asked 20 questions about Mental and physical feelings of emotional experience, and the patients determine the quality of emotion by selecting one of the options: Occasionally=1, sometimes=2, often=3, and continuously=4. The total score is multiplied by an integer of 1.25 to get the standard score.

SECONDARY OUTCOMES:
Itch perception | Baseline
  Questions regarding situations in which the itch is especially bad (multiple choice options regarding day time, daily situations); objective assessment in which respondents are asked to select answers from the choices offered as a list
Hours missing at work | Baseline and Week 2;4;8;12;16;20;24
  Approximate average hours missing at work due to itch per week from last visit.
Helpfulness of common itch therapies | Baseline and Week 2;4;8;12;16;20;24
  Questions regarding helpfulness of common itch therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhou, professor, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China